CLINICAL TRIAL: NCT04659577
Title: Attitudes of Professionals and the General Public in Israel Regarding Therapist Guided Internet Cognitive Behavioral Therapies (ICBT) to Treat Anxiety and Depression
Brief Title: Attitudes of Professionals and the General Public in Israel Regarding ICBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: Israel National Institute for Health Policy and Health Services Research (Other Government)
Responsible Party: Principal Investigator, Jonathan D. Huppert, Professor, Hebrew University of Jerusalem
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIHRP 181-15
Record Dates: First submitted 2020-05-23; First posted 2020-12-09 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Panic Disorder; Depression
MeSH Terms: conditions — Panic Disorder; Depression

STUDY DESIGN:
Intervention Model Description: All eligible people are enrolled to internet-based CBT for panic disorder or depression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- internet based CBT (Experimental): all patients will be offered active treatment via internet based CBT
  Interventions: Behavioral: ICBT for panic and depression

INTERVENTIONS:
Behavioral: ICBT for panic and depression — The most known type of CBT for treating PD consists of two major strategies: cognitive restructuring, and interoceptive and structured exposure to bodily sensations that have become associated with panic attacks. As for depression, the most known type of CBT for treating depression consists of two major strategies: cognitive restructuring, the relationship between thoughts and feelings, behavioural activation, sleep hygiene and relaxation. Each ICBT program includes six modules, containing psychoeducation, cognitive restructuring exposures, acceptance, and consolidation of gains and relapse prevention. The online modules include reading passages, worksheets, videos, and homework assignments. After completing each module participants practice related skills and complete homework assignments. The treatment is up to 16 weeks long; participants are encouraged to complete the treatment within this time period, and reminders are sent to monitor their progress
  Other Names: Internet Cognitive behavioral therapy for panic and depressive disorder.

SUMMARY:
This study examines uptake and attrition for internet based treatments for panic disorder and depression in Israel The primary benefits of this work will be a) in providing better understanding of ICBT for panic disorder and depression outcomes. Both panic and depression are heavy public health burdens, associated with a significant market potential for both therapeutic and diagnostic uses. b) In providing compatible scale to measure the working alliance during internet-based treatment.

DETAILED DESCRIPTION:
The current study examines ICBT for panic and depression in Israel. Compelling evidence regarding the efficacy of ICBT has been reported for the treatment of depression and various anxiety disorders (Mayo-Wilson & Montgomery; 2013). This the first study to examine ICBT for panic and depression in Israel. The primary focus will be on treatment outcomes (symptom reduction and improved functioning), attrition, and acceptability and comparing outcomes to previous studies of face to face and internet treatments, including on the main proposed mechanism of change; interpretation of bodily sensations via the BBSIQ. The efficacy of ICBT has been established in many studies, but is insufficient for implementation without adaptation to local cultural needs and language. We will also examine changes in healthcare utilization and costs according to the results.

For the full programs of the current study see: https://www.iterapi.se/sites/icbt_israel and https://www.iterapi.se/sites/depression_israel/

The limited role of the therapist in ICBT is mainly to allow greater scaling. a second goal of the current study is to fill this gap by examining different aspects of the alliance with treatment outcomes and attrition using a newly developed self-report measure, the Internet Patient Experiences and Attunement Responsiveness (I-PEAR). We propose that the I-PEAR and its subscales (I-PEAR program; hereafter I-PEARp, I-PEAR therapist; hereafter I-PEARt; and Therapist-rated I-PEAR; hereafter thI-PEAR) will explain more variance of the outcome and dropouts than traditional scales (i.e., WAI-6, WAI-T). In the current study we examined the relationship between the alliance measures to treatment outcomes and attrition. Alll secondary measures will be examined in terms of change and how their change is related to change in symptoms (PDSS, ASI, MI in panic, PHQ, HAM-D in depression). These analyses include changes in attachment, insight, and emotions. Research is limited about the role of insight in panic disorder, therefore another secondary aim of this study is to examine the role of clinical (i.e., SAIQ and SAI) and cognitive insight (i.e., BCIS and BABS) in panic disorder, if they change and their relationship to symptom severity (i.e., PDSS, ASI, MI), symptom change, and correlates (e.g., cognitive flexibility, metacognition, jumping to conclusions, and implicit theories). Secondary studies will examine changes in self-criticism, emotion preferences and goals, sexual functioning, and curiosity and their relationship to outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Principal DSM-5 diagnosis of panic disorder or depression
* aged 18 years or older;
* if on medications for panic or depression, the dosage has to remain constant for 2 months prior to the start of treatment and cannot be increased during treatment;
* the participant must have access to the internet and be willing to use it -

Exclusion Criteria:

* substance abuse or dependence within the last 6 months;
* active suicide potential within the last 6 months;
* any current or history of psychosis or bipolar I disorder
* currently in weekly or biweekly psychotherapy
* history of a complete course of panic or depression focused CBT

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Panic Disorder Severity Scale: Independent Evaluator Version (for panic disorder) | Weekly during treatment from pre treatment to post treatment, up to 6 months apart
  measure of a severity of panic disorder assessed by an independent evaluator. Only administered to panic patients. It is comprised of 7 items that are scored from 0-4, with a total scale score ranging from 0-28. Higher scores mean more severe panic disorder symptoms.
Change in Panic Disorder Severity Scale: Independent Evaluator Version (for panic disorder) | Baseline and 1 year follow-up
  measure of a severity of panic disorder assessed by an independent evaluator. Only administered to panic patients. It is comprised of 7 items that are scored from 0-4, with a total scale score ranging from 0-28. Higher scores mean more severe panic disorder symptoms.
Change in Hamilton Depression Scale- 17 item adjusted version | Baseline and post treatment, up to 6 months apart
  Independent evaluator measure of depression severity, higher score is more severe symptoms. total score is sum of the items, ranging from 0-52
Change in Hamilton Depression Scale- 17 item adjusted version | Baseline and 1 year follow-up
  Independent evaluator measure of depression severity, higher score is more severe symptoms.total score is sum of the items, ranging from 0-52

SECONDARY OUTCOMES:
Change in Panic disorder severity scale - self report version | Baseline and 1 year followup
  a self-report measure of panic disorder severity. Only administered to panic patients. It consists of 7 items that are scored from 0-4, with a total scale score ranging from 0-28. Higher scores mean more severe panic disorder symptoms.
Change in Panic disorder severity scale - self report version | weekly during treatment from pre treatment to post treatment, up to 6 months apart
  a self-report measure of panic disorder severity. Only administered to panic patients. It consists of 7 items that are scored from 0-4, with a total scale score ranging from 0-28. Higher scores mean more severe panic disorder symptoms.
Change in Physicians Health Questionnaire (PHQ-9) | Weekly during treatment from pre treatment to post treatment, up to 6 months apart
  A self report measure of depression- depression sample only, higher score is more severe symptoms, total scores are sums of items, ranging from 0-27.
Change in Physicians Health Questionnaire (PHQ-9) | Baseline and 1 year followup
  A self report measure of depression- depression sample only, higher score is more severe symptoms.total scores are sums of items, ranging from 0-27.
Change in Internet Patient's Experience of Attunement and Responsiveness scale (I-PEAR) | Baseline and after each module during treatment from pre treatment to post treatment
  This is an alliance scale in internet based treatment related the program and the therapist, it has been used as average between 1-5, higher score is better alliance,
Change in Anxiety Sensitivity Index (ASI) | Baseline and 1 year follow-up
  The ASI-3 is an 18-item self-report measure that measures beliefs regarding panic related bodily sensations. It will be used as a total score, which ranges from 0-72. Higher scores mean more severe anxiety sensitivity.
Change in Anxiety Sensitivity Index (ASI) | Weekly change during treatment from pre treatment to post treatment, up to 6 months apart
  The ASI-3 is an 18-item self-report measure that measures beliefs regarding panic related bodily sensations. It will be used as a total score, which ranges from 0-72. Higher scores mean more severe anxiety sensitivity.
Change in Mobility Inventory (MI) | Baseline and 1 year follow-up
  The Mobility Inventory is a self report measure of agoraphobic avoidance in which patients are asked to rate how much they avoid 26 situations on a 1-5 scale twice, once when alone and a second time when accompanied. The average score of all times will be used, which will range from 1-5. Higher total score means higher avoidance of situations. Only administered to panic patients.
Change in Mobility Inventory (MI) | Weekly change during treatment from pre treatment to post treatment, up to 6 months apart
  The Mobility Inventory is a self report measure of agoraphobic avoidance in which patients are asked to rate how much they avoid 26 situations on a 1-5 scale twice, once when alone and a second time when accompanied. The average score of all times will be used, which will range from 1-5. Higher total score means higher avoidance of situations. Only administered to panic patients.
Change in Depression Anxiety Stress Scales (DASS-21) | After each module during treatment from pre treatment to post treatment, up to 6 months apart
  A self-report measure of depression, anxiety and stress, with each subscale ranging from 0-28. for depression sample only
Change in Depression Anxiety Stress Scales (DASS-21) | Baseline and 1 year follow-up
  A self-report measure of depression, anxiety and stress, with each subscale ranging from 0-28. for depression sample only
Change in Brown Assessment of Beliefs Scale (BABS) | Baseline and post treatment, up to 6 months apart
  this is an independent evaluator measure of insight. Consists of 7 items that are rated on a scale 0-4. Higher score is worse insight, only administered to panic patients
Change in Brown Assessment of Beliefs Scale (BABS) | Baseline and 1 year follow-up
  this is an independent evaluator measure of insight. Consists of 7 items that are rated on a scale 0-4. Higher score is worse insight, only administered to panic patients
Change in Scale for the Assessment of Insight (SAI) | Baseline and post treatment, up to 6 months apart
  this is an independent evaluator measure of clinical insight. Consists of 4 items that are rated on a scale 0-2. Higher score is better insight, only administered to panic patients
Change in Scale for the Assessment of Insight (SAI) | Baseline and 1 year follow-up
  this is an independent evaluator measure of clinical insight. Consists of 4 items that are rated on a scale 0-2. Higher score is better insight, only administered to panic patients
Change in The Pittsburgh Sleep Quality Index (PSQI) | Baseline and post treatment, up to 6 months apart
  This is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, higher score is worse sleep, adminstered only to the depression sample
Change in The Pittsburgh Sleep Quality Index (PSQI) | Baseline and 1 year follow-up
  This is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, higher score is worse sleep, adminstered only to the depression sample
Change in The Sheehan Disability Scale (SDS) | Baseline and post treatment, up to 6 months apart
  this a self-report measure of disability due to an illness or health problem in work/school, social life/leisure activities, and family life/home. It includes 3 items that are rated on a scale 0-10. Higher score indicates worse disability and impairment.
Change in The Sheehan Disability Scale (SDS) | Baseline and 1 year follow-up
  this a self-report measure of disability due to an illness or health problem in work/school, social life/leisure activities, and family life/home. It includes 3 items that are rated on a scale 0-10. Higher score indicates worse disability and impairment.
Change in Self-Appraisal of Illness Questionnaire (SAIQ) | Baseline and post treatment, up to 6 months apart
  this is a self-report measure that assess clinical insight, administered only to the panic sample. It consists of 17 items that are rates on a scale 0-3. Higher scores means worse clinical insight.
Change in Self-Appraisal of Illness Questionnaire (SAIQ) | Baseline and 1 year follow-up
  this is a self-report measure that assess clinical insight, administered only to the panic sample. It consists of 17 items that are rates on a scale 0-3. Higher scores means worse clinical insight.
Change in Beck Cognitive Insight Scale (BCIS) | Baseline and 1 year follow-up
  this is a self-reported measure that assess cognitive insight, administered only to the panic sample. It consists of 15 items that are rates on a scale 0-3. Higher score means better cognitive insight.
Change in Beck Cognitive Insight Scale (BCIS) | After each module during treatment from pre treatment to post treatment, up to 6 months apart
  this is a self-reported measure that assess cognitive insight, administered only to the panic sample. It consists of 15 items that are rates on a scale 0-3. Higher score means better cognitive insight.
Change in Cognitive Flexibility Inventory (CFI) | Baseline and post treatment, up to 6 months apart
  this is a self-reported measure that assess aspects of cognitive flexibility, administered only to the panic sample. It consists of 20 items that are rated on a scale 1-7. Higher score means greater cognitive flexibility.
Change in Cognitive Flexibility Inventory (CFI) | Baseline and 1 year follow-up
  this is a self-reported measure that assess aspects of cognitive flexibility, administered only to the panic sample. It consists of 20 items that are rated on a scale 1-7. Higher score means greater cognitive flexibility.
Change in Metacognition Questionnaire - 30 item version (MCQ-30) | Baseline and post treatment, up to 6 months apart
  is a self-reported measure that assess metacognition, administered only to the panic sample. The MCQ consists of 30 items that are rated on a scale 1-4. Higher score indicated higher level of unhelpful metacognitions.
Change in Metacognition Questionnaire - 30 item version (MCQ-30) | Baseline and 1 year follow-up
  is a self-reported measure that assess metacognition, administered only to the panic sample. The MCQ consists of 30 items that are rated on a scale 1-4. Higher score indicated higher level of unhelpful metacognitions.
Change in Beck Depression Inventory -21 (BDI-21) | Baseline and post treatment, up to 6 months apart
  This is a self-report measure that assess depression, 21 items, administered only to depression sample, score ranges 0-63, higher is more severe.
Change in Beck Depression Inventory -21 (BDI-21) | Baseline and 1 year follow-up
  This is a self-report measure that assess depression, 21 items, administered only to depression sample, score ranges 0-63, higher is more severe.
Change in Implicit Theories of Emotion (TOE) | Baseline and 1 year follow-up
  Thisis a self-reported scale to measure beliefs about the fixed versus malleable nature of anxiety, administered only to the panic sample. The TOE consists of 4 items that are rates on a scale 1-5. Higher score indicates that the individual views anxiety as being relatively malleable and controllable.
Change in Implicit Theories of Emotion (TOE) | After each module during treatment from pre treatment to post treatment, up to 6 months apart
  This is a self-reported scale to measure beliefs about the fixed versus malleable nature of anxiety, administered only to the panic sample. The TOE consists of 4 items that are rates on a scale 1-5. Higher score indicates that the individual views anxiety as being relatively malleable and controllable.
Change in Implicit Theories of Thoughts (TOT) | Baseline and 1 year follow-up
  This is a self-reported scale measure beliefs about the nature of thoughts, administered only to the panic sample.The TOT consists of 4 items that are rates on a scale 1-5. Higher score indicates that the individual views thoughts as being relatively malleable and controllable.
Change in Implicit Theories of Thoughts (TOT) | After each module during treatment from pre treatment to post treatment, up to 6 months apart
  This is a self-reported scale measure beliefs about the nature of thoughts, administered only to the panic sample.The TOT consists of 4 items that are rates on a scale 1-5. Higher score indicates that the individual views thoughts as being relatively malleable and controllable.
Change in Brief Body Sensations Interpretations Questionnaire (BBSIQ) | Baseline and post treatment, up to 6 months apart
  This is a self-reported scale to measure body sensations interpretations, administered only to the panic sample. The BBSIQ includes 14 items, higher score means more negative explanation of body sensations.
Change in Brief Body Sensations Interpretations Questionnaire (BBSIQ) | Baseline and 1 year follow-up
  This is a self-reported scale to measure body sensations interpretations, administered only to the panic sample. The BBSIQ includes 14 items, higher score means more negative explanation of body sensations.
Change in Five-Dimensional Curiosity Scale (5DC) | Baseline and post treatment, up to 6 months apart
  The DCS-5 is a self-report measure that measures 5 dimensions of curiosity via 25 items which are rated on a 1-7 scale. The total score of all 25 (ranging from 25-175) items and 5 subscales (each ranging from 5-35) will be used for this study. Higher scores reflect higher curiosity. Administered only to the panic sample.
Change in Five-Dimensional Curiosity Scale (5DC) | Baseline and 1 year follow-up
  The DCS-5 is a self-report measure that measures 5 dimensions of curiosity via 25 items which are rated on a 1-7 scale. The total score of all 25 (ranging from 25-175) items and 5 subscales (each ranging from 5-35) will be used for this study. Higher scores reflect higher curiosity. Administered only to the panic sample.
Change in The five-level EuroQol five-dimensional questionnaire (EQ-5D-5L) | Baseline and post treatment, up to 6 months apart
  This is a self-reported measure of health related quality of life. It consists of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression). Higher score means worse functioning in these dimensions.
Change in The five-level EuroQol five-dimensional questionnaire (EQ-5D-5L) | Baseline and 1 year follow-up
  This is a self-reported measure of health related quality of life. It consists of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression). Higher score means worse functioning in these dimensions.
Change in Work and Social Adjustment Scale (WSAS) | Baseline and post treatment, up to 6 months apart
  This is a self-reported measure of functional impairment. It includes 5 items that are rated on a scale 0-8. Measured as total score ranging 0-40. Higher score means worse functional impairment.
Change in Work and Social Adjustment Scale (WSAS) | Baseline and 1 year follow-up
  This is a self-reported measure of functional impairment. It includes 5 items that are rated on a scale 0-8. Measured as total score ranging 0-40. Higher score means worse functional impairment.
Change in Working Alliance Inventory (WAI-6) | Baseline and post treatment, up to 6 months apart
  This is a self-reported measure of therapeutic alliance, total score is average of the items, ranging from 1-7
Change in The Experiences in Close Relationship Scale (ECR-S) | Baseline and post treatment, up to 6 months apart
  The ECR-s is a brief self report instrument that measures both anxious and avoidance adult attachment styles. The two scales each contain 6 items rated on a 1-7 scale that are averages for each subscale, ranging from 1-7. Higher score indicates an insecure adult attachment orientation.
Change in The Experiences in Close Relationship Scale (ECR-S) | Baseline and 1 year follow-up
  The ECR-s is a brief self report instrument that measures both anxious and avoidance adult attachment styles. The two scales each contain 6 items rated on a 1-7 scale that are averages for each subscale, ranging from 1-7. Higher score indicates an insecure adult attachment orientation.
Change in The Agoraphobic Cognitions Questionnaire (ACQ) | Baseline and post treatment, up to 6 months apart
  This is a self-reported scale to measure agoraphobia cognitions, administered only to the panic sample. It consists of 15 items that are rates on a scale 1-5. Higher score indicates worse dysfunctional cognitions in relation to potential catastrophic consequences arising from panic or anxiety.
Change in The Agoraphobic Cognitions Questionnaire (ACQ) | Baseline and 1 year follow-up
  This is a self-reported scale to measure agoraphobia cognitions, administered only to the panic sample. It consists of 15 items that are rates on a scale 1-5. Higher score indicates worse dysfunctional cognitions in relation to potential catastrophic consequences arising from panic or anxiety.
Change in Social Support Questionnaire (SSQ6) | Baseline and post treatment, up to 6 months apart
  This is a self-reported measure of social support. The SSQ6 includes 6 items. The overall support score is calculated by taking an average scores across the 27 items. Higher score indicates more optimism about life, higher prevalence of negative life events and illness.Scoring is as follows:
  1. Add the total number of people for all 27 items (questions). (Max. is 243). Divide by 27 for average item score.
  2. Add the total satisfaction scores for all 27 items (questions). (Max is 162). Divide by 27 for average item score. This gives you SSQ Satisfaction score or SSQS.
  3. Finally, you can average the above for the total number of people that are family members - this results in the SSQ family score. Participants indicate the number of people available to provide support in each of 6 areas and then rate the overall level of satisfaction with the supp
Change in Acceptability Scale for internet Therapy (ASIT) | Baseline and post treatment, up to 6 months apart
  This is a self-reported measure of acceptance and readiness to receive internet treatment, It consists of 19 items that are rates on a scale 1-5, total sum is ranges 1- 95, Higher score indicates more acceptability.
Change in Acceptability Scale for internet Therapy (ASIT) | Baseline and 1 year follow-up
  This is a self-reported measure of acceptance and readiness to receive internet treatment, It consists of 19 items that are rates on a scale 1-5, total sum is ranges 1- 95, Higher score indicates more acceptability.
Change in Emotional Goals Questionnaire. | Baseline and post treatment, up to 6 months apart
  This is a self-reported measure of emotional goals. is a self-reported measure of emotional goals. The measure assesses emotional preferences ro feel unpleasant emotions of (eg., depression, anxiety, etc) and beliefs about the fixed versus malleable nature of anxiety. Higher score indicates higher ability and willingness to feel unpleasant emotions and that the individual views anxiety as being relatively malleable and controllable.

OTHER OUTCOMES:
Change in questionnaire of Implicit Association Test (qIAT) for Experiences in Close Relationship Scale-Short | Baseline and post treatment, up to 6 months apart
  The Questionnaire-based Implicit Association Test (qIAT) associated with the conventional self-concept IAT, and it enables an indirect assessment that is based on the items of standard self-reports. The current qIAT is related the ECR for attachment and administered separetely for anxious (4 items) for avoidant (4 items).
Change in Depressive Experience Questionnaire (DEQ) | After each module from pre treatment to post treatment, up to 6 months apart
  A self -report scale about self critisism which is related to depressive symptoms, 11 items, higher is more severe, administered to depression sample only.
Change in Depressive Experience Questionnaire (DEQ) | Baseline and 1 year follow-up
  A self -report scale about self critisism which is related to depressive symptoms,11 items, ranging 1-7 higher is more severe, administered to depression sample only.
Change in Distressing Thoughts | Baseline and post treatment, up to 6 months apart
  A task about distressing thoughts. Participants have to imagine distressing situation and then after 4 minutes to describe their thoughts.
Change in Distressing Thoughts | Baseline and 1 year follow-up
  A task about distressing thoughts. Participants have to imagine distressing situation and then after 4 minutes to describe their thoughts.
Change in Current Emotion | Baseline and post treatment, up to 6 months apart
  A self report about current emotions, more sad emotion is related to depression, 8 items, total score is average ranging 1-7,administered to depression sample only . administered to depression sample only
Change in Current Emotion | Baseline and 1 year follow-up
  A self report about current emotions, more sad emotion is related to depression, 8 items, total score is average ranging 1-7,administered to depression sample only . administered to depression sample only
Change in Emotional Preferences | Baseline and post treatment, up to 6 months apart
  A self report about emotional preferences, more sad emotion is related to depression, 10 items, total score is average ranging 1-7, administered to depression sample only
Change in Emotional Preferences | Baseline and 1 year follow-up
  A self report about emotional preferences, more sad emotion is related to depression, 10 items, total score is average ranging 1-7, administered to depression sample only
Change in Emotional Preferences Task | Baseline and post treatment, up to 6 months apart
  A task about emotional preferences, in this task participants choose which photo they prefer to see. administered to depression sample only
Change in State-Reappraisal Inventory (SRI) | after each module during treatment from pre treatment to post treatment, up to 6 months apart
  A self report scale about state reappraisal, related to self regulation, 12 items, total score is avarge ranging 1-5, lower score related to more ability to reappraisal and self regulation. administered in depression sample only.